CLINICAL TRIAL: NCT03388554
Title: To Investigate the Effects of Transcranial Direct Current Stimulation on Auditory Hallucination, Insight, Neurocognitive Function, Heart Rate Variability, Psychosocial Functioning and Quality of Life in Patients With Schizophrenia
Brief Title: The Effects of tDCS on Auditory Hallucination, Insight, Neurocognitive Function and HRV in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Head of Laboratory of Psychophysiology, Department of Psychiatry, Principal Investigator, Attending Psychiatrist, Assistant Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-103-03-002-2
Record Dates: First submitted 2017-12-24; First posted 2018-01-03 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Auditory Hallucination, Verbal; Neurocognitive Dysfunction; Autonomic Imbalance; Psychosocial Impairment; Quality of Life
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations; Cognition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Direct current (DC) generated by a DC stimulator (Eldith DC stimulator: www. neuroconn.de/dc-stimulator_plus_en/) was bilaterally delivered through a pair of saline-soaked surface sponge electrodes (35 square centimeter). The anode was placed with the middle of the electrode over a point midway between F3 and FP1 (left dorsolateral prefrontal cortex and left prefrontal cortex). The cathode was located over a point midway between T3 and P3 (left temporo-parietal junction). Stimulation was applied at an intensity of 2 mA for 20 min, twice-daily on 5 consecutive weekdays. The twice daily sessions were separated by at least 3 hours.
Who Masked: Participant, Outcomes Assessor
Masking Description: In sham stimulation, the current was turned on for 30 sec and then ramped down to 0 mA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Direct current (DC) generated by a DC stimulator (Eldith DC stimulator: www. neuroconn.de/dc-stimulator_plus_en/) was bilaterally delivered through a pair of saline-soaked surface sponge electrodes (35 square centimeter). The anode was placed with the middle of the electrode over a point midway between F3 and FP1 (left dorsolateral prefrontal cortex and left prefrontal cortex). The cathode was located over a point midway between T3 and P3 (left temporo-parietal junction). Stimulation was applied at an intensity of 2 mA for 20 min, twice-daily on 5 consecutive weekdays. The twice daily sessions were separated by at least 3 hours. All patients in the active tDCS group were maintained on their antipsychotic medications throughout the study period.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): In sham stimulation, the current was turned on for 30 sec and then ramped down to 0 mA. All patients in the sham tDCS group were maintained on their antipsychotic medications throughout the study period.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS

SUMMARY:
The study aimed to investigate whether transcranial direct current stimulation could modify auditory hallucination, insight, neurocognitive function, heart rate variability, psychosocial functioning and quality of life in patients with schizophrenia.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS), a novel, non-invasive and safe neuro-modulating technique, has been developed as a new therapeutic option for neuropsychiatric disorders. It encompasses the induction of a relatively weak constant current flow through the cerebral cortex via scalp electrodes. Dependent on stimulation polarity, this results in a modulation of cortical excitability and spontaneous neural activity. The technique was established in the 1950s and 1960s primarily in animals. In these early studies it was shown that subthreshold DC stimulation increases spontaneous neuronal activity if the anode is placed above or within the cortex, while exposure to cathodal polarity results in reduced activity. This is caused by a subthreshold membrane depolarization by anodal and a hyperpolarization by cathodal stimulation. It was demonstrated in humans that the after-effects of tDCS depend on modifications of NMDA receptor-efficacy. The after-effects of tDCS are blocked by the NMDA receptor antagonist dextromethorphan, and prolonged by the partial NMDA receptor-agonist D-cycloserine. This tDCS polarity-dependent alteration of NMDA receptor function seems to be initiated by the respective membrane potential shift and probably by the accompanying cortical activity modification,because it is prevented by the sodium channel blocker carbamazepine. Intraneuronal calcium concentration also contributes, because calcium channel antagonists eliminate the excitability-enhancing aftereffects of anodal tDCS. Recently, tDCS has been found to improve psychopathological symptoms (auditory hallucination in particular), cognitive deficits and insight of schizophrenia and also strengthen cardiac autonomic function in healthy subjects. Further replication studies are needed.

The study aimed to investigate whether transcranial direct current stimulation could modify auditory hallucination, insight, neurocognitive function, heart rate variability, psychosocial functioning and quality of life in patients with schizophrenia.

Study design: randomized double-blind, sham-controlled study design.

Participants: 60 patients having a diagnosis of schizophrenia or schizoaffective with refractory auditory verbal hallucinations (defined as the persistence of daily auditory verbal hallucinations without remission in spite of antipsychotic medications at an adequate dosage for at least 3 months), aged 20-65 years.

Others: see Arms and Interventions, Eligibility Criteria or Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

- Patients who met DSM-IV-TR criteria for schizophrenia or schizoaffective disorder were included in the study. All these patients showed refractory auditory verbal hallucinations,which are defined as the persistence of daily auditory verbal hallucinations without remission in spite of antipsychotic medications at an adequate dosage for at least 3 months.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Having epilepsy, severe physical illness, any current psychiatric comorbidity or history of substance dependence.
3. Having contraindications for transcranial electrical/magnetic stimulation.
4. Having intracranial metal foreign bodies.
5. Having a history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline scores of Auditory Hallucination Rating Scale (AHRS) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  A clinician-administered rating scale to measure the severity of auditory (verbal) hallucination of the patients with schizophrenia spectrum disorder.

SECONDARY OUTCOMES:
Changes from baseline scores of Positive and Negative Syndrome Scale (PANSS) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  A clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder.
Changes from baseline scores at Personal and Social Performance scale (PSP) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  A clinician-administered rating scale to measure the psychosocial functioning of the patients with schizophrenia spectrum disorder.
Changes from baseline results of Digit span (forward and backward) | One month.
  A test to measure the capacity of working memory of the patients.
Changes from baseline results of Finger tapping test | One month.
  A neuropsychological test that examines motor functioning, specifically, motor speed and lateralized coordination.
Changes from baseline results of Continuous Performance (CPT, version 2.0) | One month.
  A neuropsychological test that examines the performance of prefrontal-mediated task.
Changes from baseline results of Wisconsin Card Sorting Test (WCST) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.
Changes from baseline results of Trail Making Test (TMT) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A neuropsychological test of visual attention and task switching.
Changes from baseline results of Tower of London test at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A neuropsychological test for the assessment of executive functioning specifically to detect deficits in planning, which may occur due to a variety of medical and neuropsychiatric conditions.
Changes from baseline heart rate variability (HRV) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  An index of autonomic functioning.
Changes from baseline scores of the brief version of questionnaire of The World Health Organization Quality of Life (WHOQOL-BREF Taiwan version) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A self-reported questionnaire to measure quality of life of the patients.
Changes from baseline scores of self-reported version of the graphic Personal and Social Performance scale (SRG-PSP) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  A self-reported graphic questionnaire to measure psychosocial functioning of the patients.
Changes from baseline scores of the abbreviated version of the Scale to Assess Unawareness in Mental Disorder in schizophrenia (SUMD) at the timepoint immediately after tDCS, at one month and three months after tDCS. | Three months.
  An expert-rating scale based on a patient interview to measure the insight of the patient.
Changes from baseline scores of the Taiwanese version of the Beck Cognitive Insight Scale (BCIS) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  Translated BCIS has two subscales including reflective attitude (R, 9 items, score range 9-36) and certain attitude (C, 6 items, score range 6-24) subscales. The higher score in R subscale indicates higher self-reflectiveness while the higher score in C subscale indicates higher self-certainty. Thus, a composite index (R-C, reflective attitude minus certain attitude, score range 3-30) of the translated BCIS represents the measurement of cogntive insight . The higher score of R-C index indicates higher cognitive insight.
Changes from baseline scores of the Taiwanese version of the Self- Appraisal of Illness Questionnaire (SAIQ) at the timepoint immediately after tDCS and at one month after tDCS. | One month.
  This scale is a self-report instrument composed of 17 items on which participants are asked to rate the extent to which they agree with each statement using a four-point Likert scale, ranging from 0, ''do not agree at all'', to 3, ''agree completely'', which varies according to the statement or questions content. SAIQ has three subscales including worry, need for treatment, and presence/outcome of illness subscales. The scores for the three subscales were summed to create a total SAIQ score (range 17-68), which is intended to represent a broad measure of insight. Lower SAIQ total scores indicate less awareness of one's psychiatric illness.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-service general hospital, Taipei, Taiwan